CLINICAL TRIAL: NCT02644473
Title: Safety of Topical Tranexamic Acid in Total Joint Arthroplasty in High Risk Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study did not receive IRB approval, so did not start
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-5435
Record Dates: First submitted 2015-12-30; First posted 2015-12-31 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2015-12

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Stroke; Myocardial Infarction
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Stroke; Myocardial Infarction | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (Experimental): Investigators will administer topical (1.5g) TXA during total knee arthroplasty and total hip arthroplasty
  Interventions: Drug: Tranexamic Acid
- Control (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic acid
Drug: Normal saline — Control
  Arms: Control

SUMMARY:
To evaluate whether there is a difference in symptomatic thromboembolism events in the subset of patients with a history of, or risk factors for thromboembolic disease for topically applied tranexamic acid in total joint arthroplasty.

DETAILED DESCRIPTION:
Tranexamic acid (TXA) has been used successfully to stop bleeding after dental procedures, removal of tonsils, prostate surgery, heavy menstrual bleeding, and eye injuries, as well as in patients with hemophilia. Intravenous TXA has also been shown to reduce blood loss, reduce transfusion requirements, and decrease length of stay for patients undergoing total knee arthroplasty and total hip arthroplasty. These benefits occur without increasing risks of thromboembolism events such as pulmonary embolism, deep venous thrombosis, myocardial infarctions, and cerebrovascular events in patients without history of, or risk factors for thromboembolic disease. Topical TXA in TJA has also been demonstrated to show the above benefits without any increase risks, as well as systemic absorption of the medication that is below the effective therapeutic plasma concentration.

Preliminary retrospective studies has demonstrated that IV TXA to be safe and effective in patients with risk factors for thromboembolic events and patients with American Society of Anesthesiologists score III or IV.

Currently, there are no prospective studies on the use of either IV or topical TXA in these higher risk patients. The goal of this study is to evaluate whether there is a difference in symptomatic thromboembolism events in the subset of patients with a history of, or risk factors for thromboembolic disease for topically applied TXA in total joint arthroplasty (TJA).

ELIGIBILITY:
Inclusion Criteria:

Presence of one or more of seven risk factors for thromboembolic events - Prior DVT, PE, MI, CVA, coronary artery stent placement, CABG, or prothrombotic condition (Factor V Leiden deficiency, protein C deficiency, antiphospholipid syndrome, etc).

Exclusion Criteria:

Simultaneous bilateral, hip resurfacing, partial knee, and revision arthroplasties

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Deep Vein Thrombosis | 1 month
Pulmonary Embolism | 1 month
Stroke | 1 month
Myocardial infarction | 1 month

REFERENCES:
- [Background] Jansen AJ, Andreica S, Claeys M, D'Haese J, Camu F, Jochmans K. Use of tranexamic acid for an effective blood conservation strategy after total knee arthroplasty. Br J Anaesth. 1999 Oct;83(4):596-601. doi: 10.1093/bja/83.4.596. PMID 10673876
- [Background] McCormack PL. Tranexamic acid: a review of its use in the treatment of hyperfibrinolysis. Drugs. 2012 Mar 26;72(5):585-617. doi: 10.2165/11209070-000000000-00000. PMID 22397329
- [Background] Zhang H, Chen J, Chen F, Que W. The effect of tranexamic acid on blood loss and use of blood products in total knee arthroplasty: a meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2012 Sep;20(9):1742-52. doi: 10.1007/s00167-011-1754-z. Epub 2011 Nov 8. PMID 22065294
- [Background] Alshryda S, Mason J, Sarda P, Nargol A, Cooke N, Ahmad H, Tang S, Logishetty R, Vaghela M, McPartlin L, Hungin AP. Topical (intra-articular) tranexamic acid reduces blood loss and transfusion rates following total hip replacement: a randomized controlled trial (TRANX-H). J Bone Joint Surg Am. 2013 Nov 6;95(21):1969-74. doi: 10.2106/JBJS.L.00908. PMID 24196467
- [Background] Huang Z, Ma J, Shen B, Pei F. Combination of intravenous and topical application of tranexamic acid in primary total knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Dec;29(12):2342-6. doi: 10.1016/j.arth.2014.05.026. Epub 2014 Jun 5. PMID 25007725
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] Whiting DR, Gillette BP, Duncan C, Smith H, Pagnano MW, Sierra RJ. Preliminary results suggest tranexamic acid is safe and effective in arthroplasty patients with severe comorbidities. Clin Orthop Relat Res. 2014 Jan;472(1):66-72. doi: 10.1007/s11999-013-3134-0. PMID 23817754
- [Background] Duncan CM, Gillette BP, Jacob AK, Sierra RJ, Sanchez-Sotelo J, Smith HM. Venous thromboembolism and mortality associated with tranexamic acid use during total hip and knee arthroplasty. J Arthroplasty. 2015 Feb;30(2):272-6. doi: 10.1016/j.arth.2014.08.022. Epub 2014 Sep 6. PMID 25257237